CLINICAL TRIAL: NCT01156376
Title: Determination of the Oral Irritation and Sensitization Potential of Two Experimental Potassium Oxalate Containing Mouthrinses
Brief Title: Oral Irritation Study of Two Experimental Mouthrinses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KOXDHY0003
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Oral Manifestations
MeSH Terms: conditions — Oral Manifestations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PO-019 (Experimental): Formula 12027-019 Mouthwash
  Interventions: Device: Potassium Oxalate without Fluoride
- PO-020 (Experimental): Formula 12027-020 Mouthwash
  Interventions: Device: Potassium Oxalate with Fluoride
- PO-116-A (Active Comparator): Cool Mint Listerine
  Interventions: Device: Active Comparator PO-116-A

INTERVENTIONS:
Device: Potassium Oxalate without Fluoride — 1.40% Potassium Oxalate Sensitive Mouthwash without fluoride - Rinse with 10ml for 60 seconds, four times daily successively at 1 hour intervals for five days
  Other Names: Formula 12027-019
  Arms: PO-019
Device: Potassium Oxalate with Fluoride — 1.40% Potassium Oxalate Sensitive Mouthwash with fluoride - Rinse with 20ml for 60 seconds, four times daily successively at 1 hour intervals for five days
  Other Names: Formula 12027-020
  Arms: PO-020
Device: Active Comparator PO-116-A — Rinse with comparator mouthwash 20ml for 30 seconds, four times daily successively at 1 hour intervals for five days
  Other Names: Cool Mint Listerine
  Arms: PO-116-A

SUMMARY:
This study is 25 days long. People participating in this study will be asked to brush their teeth two times a day. People will be assigned to a mouthwash and will rinse four times a day at the site for five days. A dentist or dental hygienist will look at the mouth, teeth, tongue and gums to make sure the mouthwash does not irritate the mouth. After Day 5 of the study, people will continue to brush two times a day and will return on Day 24 to have their mouth looked at again. People without irritation in their mouth will rinse 4 times a day at the clinical site. People will return to the clinical site the next day and have a final oral exam in which the dentist or dental hygienist will look at the mouth for irritation.

DETAILED DESCRIPTION:
This is a randomized, observer-blind, single-center, supervised, controlled, parallel-designed study. Approximately 90 generally healthy adults meeting the necessary inclusion/exclusion criteria will be enrolled so that 78 subjects (26 per treatment group) would reasonably be expected to complete the study. Subjects will have their oral soft/hard tissues assessed at Screening (visit 1), Baseline (visit 2), and Days 3, 5, 24, and 25 (visits 4,6-8). During the first week of the study, subjects will be instructed to brush their teeth for one minute in their usual manner, twice daily using the provided standard fluoride toothpaste. Subjects will return for the Baseline exam and, upon qualification with entry criteria, will be assigned to one of three treatment groups. Qualified subjects will be instructed to return to the site for five consecutive days. Subjects will have four supervised rinses with their assigned mouth rinse for either 30 or 60 seconds using 10 ml or 20 ml, at subsequent one-hour intervals. During the 5 consecutive days of exposure to the assigned mouthrinse, subjects will brush their teeth using the provided fluoride-free toothpaste and soft-bristled toothbrush.

Subjects will then have an 18-day rest period (off treatment). During this time, subjects will follow their usual oral hygiene and dietary habits, using the standard fluoride toothpaste and soft toothbrush provided, and must refrain from using any unassigned oral care products. On the 19th day after completion of Day 5 (Day 24), subjects will return for an oral examination. If no pathology is present, subjects will be given a challenge treatment (four supervised rinses) and the final oral examination will be performed on Day 25.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age in good general and oral health without any known allergy to commercial dental products or cosmetics.
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Willingness to use the assigned products according to instructions, availability for appointments, and likelihood of completing the clinical trial.
* Willingness to refrain from using any breath freshener products (e.g., oral care strips, candy-type mints, sprays, chewing gums, throat lozenges, cough drops or mouthwashes), whitening products and smokeless tobacco products within one week prior to and for the duration of the study, in order to reduce alternate sources of potential irritation and sensitization.
* A minimum of 20 natural teeth.
* Absence of abnormal or severe fissured tongue, geographic tongue, or any obvious tongue abnormalities that may interfere with the assessment of oral irritation.
* Adequate oral hygiene (i.e., brush teeth daily & exhibit no signs of oral neglect).
* Absence of neglected dental health (i.e., gross calculus deposits or rampant caries based on visual examination), significant oral soft tissue pathology, systematically-related gingival enlargement or tissue damage due to ill-fitting appliances or restoration.
* Absence of orthodontic bands, appliances, bridges, extensive large restorations or removable orthodontic appliances.

Exclusion Criteria:

* Volunteers who report history or presence of kidney disorders or kidney stones, Crohn's Disease or other malabsorption syndromes.
* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthwashes.
* Physical limitations or restrictions that might preclude use of normal oral hygiene procedures (i.e., toothbrushing, mouthrinsing, etc.).
* History or current evidence of significant oral soft tissue pathology, excluding gingivitis, based on the dentist's visual examination and at the discretion of the investigator.
* Those requiring antibiotic premedication prior to dental treatment.
* Participation in a dental clinical trial involving oral care products within the past 30 days.
* Visual evidence of Moderate/Advanced Periodontitis (ADA Type III, IV).
* Women who are pregnant, nursing or plan to become pregnant during the course of the study.
* Volunteers requiring treatment with Indinavir or loop diuretics (i.e., Furosemide).
* Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial result and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial
* Any clinical history which in the opinion of the investigator could compromise the safety of the subject or the clinical parameters being assessed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, DMD, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- University Park Research Center (UPRC), Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 19292-116-A Control (Listerine®): Cool Mint® Listerine® Antiseptic Mouth Rinse (20 mL)
- 12027-019: 1.40% Potassium Oxalate Mouth Rinse without Fluoride (10 mL)
- 12027-020: 1.40% Potassium Oxalate Mouth Rinse with Fluoride (20 mL)
Period: Overall Study
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Started | 27 | 26 | 27
Completed | 26 | 26 | 23
Not Completed | 1 | 0 | 4
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020 | Total
Number analyzed (Participants) | 27 | 26 | 27 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (14.24) | 37.6 (14.29) | 51.0 (15.03) | 45.8 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 22 | 57
  Male | 7 | 11 | 5 | 23
Region of Enrollment [Number; unit: participants]
  USA | 27 | 26 | 27 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Abnormal Condition by Anatomical Site at Screening
Description: Buccal, labial and sublingual mucosae, mucobuccal fold, gingiva, tongue, hard and soft palate, uvula, oropharynx, teeth and dental restorations were examined. The dental examiner evaluated any condition as either normal or abnormal.
Time Frame: Screening
Population: Analysis was based on subjects with measurements for this variable.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  Buccal Mucosa | 0 | 0 | 0
  Labial Mucosa | 0 | 0 | 0
  Sublingual Mucosa | 0 | 0 | 0
  Mucobuccal Fold | 0 | 3.8 | 0
  Gingiva | 0 | 0 | 3.7
  Tongue | 0 | 3.8 | 3.7
  Hard/Soft Palate | 0 | 0 | 0
  Uvula/Oropharynx | 0 | 0 | 0
  Teeth | 0 | 0 | 0
  Dental Restorations | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With an Abnormal Condition by Anatomical Site at Day 1 - Baseline/Pretreatment
Description: as for outcome 1
Time Frame: Day 1 - Baseline/Pretreatment
Population: Analysis was based on subjects with measurements for this variable.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  Buccal Mucosa | 0 | 0 | 0
  Labial Mucosa | 0 | 0 | 0
  Sublingual Mucosa | 0 | 0 | 0
  Mucobuccal Fold | 0 | 0 | 0
  Gingiva | 0 | 0 | 0
  Tongue | 3.7 | 0 | 3.7
  Hard/Soft Palate | 0 | 0 | 0
  Uvula/Oropharynx | 0 | 0 | 0
  Teeth | 0 | 0 | 0
  Dental Restorations | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With an Abnormal Condition by Anatomical Site at Day 1 - Post-treatment
Description: as for outcome 1
Time Frame: Day 1 - Post-treatment
Population: Analysis was based on subjects with measurements for this variable.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  Buccal Mucosa | 0 | 0 | 3.8
  Labial Mucosa | 0 | 0 | 0
  Sublingual Mucosa | 0 | 0 | 0
  Mucobuccal Fold | 0 | 0 | 0
  Gingiva | 0 | 0 | 0
  Tongue | 18.5 | 0 | 7.7
  Hard/Soft Palate | 0 | 0 | 0
  Uvula/Oropharynx | 0 | 0 | 0
  Teeth | 0 | 0 | 0
  Dental Restorations | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With an Abnormal Condition by Anatomical Site at Day 3
Description: as for outcome 1
Time Frame: Day 3
Population: Analysis was based on subjects with measurements for this variable.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  Buccal Mucosa | 0 | 0 | 3.8
  Labial Mucosa | 0 | 0 | 0
  Sublingual Mucosa | 0 | 0 | 0
  Mucobuccal Fold | 0 | 0 | 0
  Gingiva | 0 | 0 | 0
  Tongue | 25.9 | 0 | 3.8
  Hard/Soft Palate | 0 | 0 | 0
  Uvula/Oropharynx | 0 | 0 | 0
  Teeth | 0 | 0 | 0
  Dental Restorations | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants With an Abnormal Condition by Anatomical Site at Day 5
Description: as for outcome 1
Time Frame: Day 5
Population: Analysis was based on subjects with measurements for this variable.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  Buccal Mucosa | 0 | 0 | 4.0
  Labial Mucosa | 0 | 0 | 0
  Sublingual Mucosa | 0 | 0 | 0
  Mucobuccal Fold | 0 | 0 | 0
  Gingiva | 0 | 0 | 0
  Tongue | 22.2 | 0 | 4.0
  Hard/Soft Palate | 0 | 0 | 0
  Uvula/Oropharynx | 0 | 0 | 0
  Teeth | 0 | 0 | 0
  Dental Restorations | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants With an Abnormal Condition by Anatomical Site at Day 24 - Pretreatment
Description: as for outcome 1
Time Frame: Day 24 - Pretreatment
Population: Analysis was based on subjects with measurements for this variable.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  Buccal Mucosa | 3.7 | 0 | 0
  Labial Mucosa | 0 | 0 | 0
  Sublingual Mucosa | 0 | 0 | 0
  Mucobuccal Fold | 0 | 0 | 0
  Gingiva | 0 | 0 | 0
  Tongue | 3.7 | 0 | 4.3
  Hard/Soft Palate | 0 | 0 | 0
  Uvula/Oropharynx | 0 | 0 | 0
  Teeth | 0 | 0 | 0
  Dental Restorations | 0 | 0 | 0

7. Primary Outcome: Percentage of Participants With an Abnormal Condition by Anatomical Site at Day 24 - Post-treatment
Description: as for outcome 1
Time Frame: Day 24 - Post-treatment
Population: Analysis was based on subjects with measurements for this variable.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  Buccal Mucosa | 0 | 0 | 0
  Labial Mucosa | 0 | 0 | 0
  Sublingual Mucosa | 0 | 0 | 0
  Mucobuccal Fold | 0 | 0 | 0
  Gingiva | 0 | 0 | 0
  Tongue | 15.4 | 0 | 4.3
  Hard/Soft Palate | 0 | 0 | 0
  Uvula/Oropharynx | 0 | 0 | 0
  Teeth | 0 | 0 | 0
  Dental Restorations | 0 | 0 | 0

8. Primary Outcome: Percentage of Participants With an Abnormal Condition by Anatomical Site at Day 25
Description: as for outcome 1
Time Frame: Day 25
Population: Analysis was based on subjects with measurements for this variable.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  Buccal Mucosa | 0 | 0 | 0
  Labial Mucosa | 0 | 0 | 0
  Sublingual Mucosa | 0 | 0 | 0
  Mucobuccal Fold | 0 | 0 | 0
  Gingiva | 0 | 0 | 0
  Tongue | 0 | 0 | 4.3
  Hard/Soft Palate | 0 | 0 | 0
  Uvula/Oropharynx | 0 | 0 | 0
  Teeth | 0 | 0 | 0
  Dental Restorations | 0 | 0 | 0

9. Primary Outcome: Percentage of Subjects in Irritation Score Category for Buccal Mucosa at Screening
Description: The dental examiner rated the irritation/inflammation on the soft tissues using a scale where 0=none (normal), 1=erythema plus slight edema (mild), 2=moderate erythema and/or edema (beginning of tissue breakdown or sloughing) (moderate), 3=severe inflammation/irritation (definite blistering, ulceration, or epithelial sloughing) (severe).
Time Frame: Screening
Population: Analysis was based on the Full Analysis Set, defined as all randomized participants who used the investigational product. No imputations were made for missing data.
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

10. Primary Outcome: Percentage of Subjects in Irritation Score Category for Labial Mucosa at Screening
Description: as for outcome 9
Time Frame: Screening
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

11. Primary Outcome: Percentage of Subjects in Irritation Score Category for Sublingual Mucosa at Screening
Description: as for outcome 9
Time Frame: Screening
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

12. Primary Outcome: Percentage of Subjects in Irritation Score Category for Mucobuccal Fold at Screening
Description: as for outcome 9
Time Frame: Screening
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 96.2 | 100
  Mild | 0 | 3.8 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

13. Primary Outcome: Percentage of Subjects in Irritation Score Category for Gingiva at Screening
Description: as for outcome 9
Time Frame: Screening
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

14. Primary Outcome: Percentage of Subjects in Irritation Score Category for Tongue at Screening
Description: as for outcome 9
Time Frame: Screening
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 96.2 | 100
  Mild | 0 | 3.8 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

15. Primary Outcome: Percentage of Subjects in Irritation Score Category for Hard/Soft Palate at Screening
Description: as for outcome 9
Time Frame: Screening
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

16. Primary Outcome: Percentage of Subjects in Irritation Score Category for Uvula/Oropharynx at Screening
Description: as for outcome 9
Time Frame: Screening
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

17. Primary Outcome: Percentage of Subjects in Irritation Score Category for Buccal Mucosa at Day 1 - Baseline/Pretreatment
Description: as for outcome 9
Time Frame: Day 1 - Baseline/Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

18. Primary Outcome: Percentage of Subjects in Irritation Score Category for Labial Mucosa at Day 1 - Baseline/Pretreatment
Description: as for outcome 9
Time Frame: Day 1 - Baseline/Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

19. Primary Outcome: Percentage of Subjects in Irritation Score Category for Sublingual Mucosa at Day 1 - Baseline/Pretreatment
Description: as for outcome 9
Time Frame: Day 1 - Baseline/Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

20. Primary Outcome: Percentage of Subjects in Irritation Score Category for Mucobuccal Fold at Day 1 - Baseline/Pretreatment
Description: as for outcome 9
Time Frame: Day 1 - Baseline/Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

21. Primary Outcome: Percentage of Subjects in Irritation Score Category for Gingiva at Day 1 - Baseline/Pretreatment
Description: as for outcome 9
Time Frame: Day 1 - Baseline/Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

22. Primary Outcome: Percentage of Subjects in Irritation Score Category for Tongue at Day 1 - Baseline/Pretreatment
Description: as for outcome 9
Time Frame: Day 1 - Baseline/Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 96.3 | 100 | 100
  Mild | 3.7 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

23. Primary Outcome: Percentage of Subjects in Irritation Score Category for Hard/Soft Palate at Day 1 - Baseline/Pretreatment
Description: as for outcome 9
Time Frame: Day 1 - Baseline/Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

24. Primary Outcome: Percentage of Subjects in Irritation Score Category for Uvula/Oropharynx at Day 1 - Baseline/Pretreatment
Description: as for outcome 9
Time Frame: Day 1 - Baseline/Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 27
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

25. Primary Outcome: Percentage of Subjects in Irritation Score Category for Buccal Mucosa at Day 1 - Post-treatment
Description: as for outcome 9
Time Frame: Day 1 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 96.2
  Mild | 0 | 0 | 3.8
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

26. Primary Outcome: Percentage of Subjects in Irritation Score Category for Labial Mucosa at Day 1 - Post-treatment
Description: as for outcome 9
Time Frame: Day 1 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

27. Primary Outcome: Percentage of Subjects in Irritation Score Category for Sublingual Mucosa at Day 1 - Post-treatment
Description: as for outcome 9
Time Frame: Day 1 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

28. Primary Outcome: Percentage of Subjects in Irritation Score Category for Mucobuccal Fold at Day 1 - Post-treatment
Description: as for outcome 9
Time Frame: Day 1 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

29. Primary Outcome: Percentage of Subjects in Irritation Score Category for Gingiva at Day 1 - Post-treatment
Description: as for outcome 9
Time Frame: Day 1 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

30. Primary Outcome: Percentage of Subjects in Irritation Score Category for Tongue at Day 1 - Post-treatment
Description: as for outcome 9
Time Frame: Day 1 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 96.3 | 100 | 96.2
  Mild | 3.7 | 0 | 3.8
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

31. Primary Outcome: Percentage of Subjects in Irritation Score Category for Hard/Soft Palate at Day 1 - Post-treatment
Description: as for outcome 9
Time Frame: Day 1 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

32. Primary Outcome: Percentage of Subjects in Irritation Score Category for Uvula/Oropharynx at Day 1 - Post-treatment
Description: as for outcome 9
Time Frame: Day 1 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

33. Primary Outcome: Percentage of Subjects in Irritation Score Category for Buccal Mucosa at Day 3
Description: as for outcome 9
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 96.2
  Mild | 0 | 0 | 3.8
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

34. Primary Outcome: Percentage of Subjects in Irritation Score Category for Labial Mucosa at Day 3
Description: as for outcome 9
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

35. Primary Outcome: Percentage of Subjects in Irritation Score Category for Sublingual Mucosa at Day 3
Description: as for outcome 9
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

36. Primary Outcome: Percentage of Subjects in Irritation Score Category for Mucobuccal Fold at Day 3
Description: as for outcome 9
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

37. Primary Outcome: Percentage of Subjects in Irritation Score Category for Gingiva at Day 3
Description: as for outcome 9
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

38. Primary Outcome: Percentage of Subjects in Irritation Score Category for Tongue at Day 3
Description: as for outcome 9
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

39. Primary Outcome: Percentage of Subjects in Irritation Score Category for Hard/Soft Palate at Day 3
Description: as for outcome 9
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

40. Primary Outcome: Percentage of Subjects in Irritation Score Category for Uvula/Oropharynx at Day 3
Description: as for outcome 9
Time Frame: Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 26
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

41. Primary Outcome: Percentage of Subjects in Irritation Score Category for Buccal Mucosa at Day 5
Description: as for outcome 9
Time Frame: Day 5
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  None | 100 | 100 | 96.0
  Mild | 0 | 0 | 4.0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

42. Primary Outcome: Percentage of Subjects in Irritation Score Category for Labial Mucosa at Day 5
Description: as for outcome 9
Time Frame: Day 5
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

43. Primary Outcome: Percentage of Subjects in Irritation Score Category for Sublingual Mucosa at Day 5
Description: as for outcome 9
Time Frame: Day 5
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

44. Primary Outcome: Percentage of Subjects in Irritation Score Category for Mucobuccal Fold at Day 5
Description: as for outcome 9
Time Frame: Day 5
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

45. Primary Outcome: Percentage of Subjects in Irritation Score Category for Gingiva at Day 5
Description: as for outcome 9
Time Frame: Day 5
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

46. Primary Outcome: Percentage of Subjects in Irritation Score Category for Tongue at Day 5
Description: as for outcome 9
Time Frame: Day 5
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

47. Primary Outcome: Percentage of Subjects in Irritation Score Category for Hard/Soft Palate at Day 5
Description: as for outcome 9
Time Frame: Day 5
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

48. Primary Outcome: Percentage of Subjects in Irritation Score Category for Uvula/Oropharynx at Day 5
Description: as for outcome 9
Time Frame: Day 5
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 25
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

49. Primary Outcome: Percentage of Subjects in Irritation Score Category for Buccal Mucosa at Day 24 - Pretreatment
Description: as for outcome 9
Time Frame: Day 24 - Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  None | 96.3 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 3.7 | 0 | 0
  Severe | 0 | 0 | 0

50. Primary Outcome: Percentage of Subjects in Irritation Score Category for Labial Mucosa at Day 24 - Pretreatment
Description: as for outcome 9
Time Frame: Day 24 - Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

51. Primary Outcome: Percentage of Subjects in Irritation Score Category for Sublingual Mucosa at Day 24 - Pretreatment
Description: as for outcome 9
Time Frame: Day 24 - Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

52. Primary Outcome: Percentage of Subjects in Irritation Score Category for Mucobuccal Fold at Day 24 - Pretreatment
Description: as for outcome 9
Time Frame: Day 24 - Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

53. Primary Outcome: Percentage of Subjects in Irritation Score Category for Gingiva at Day 24 - Pretreatment
Description: as for outcome 9
Time Frame: Day 24 - Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

54. Primary Outcome: Percentage of Subjects in Irritation Score Category for Tongue at Day 24 - Pretreatment
Description: as for outcome 9
Time Frame: Day 24 - Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

55. Primary Outcome: Percentage of Subjects in Irritation Score Category for Hard/Soft Palate at Day 24 - Pretreatment
Description: as for outcome 9
Time Frame: Day 24 - Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

56. Primary Outcome: Percentage of Subjects in Irritation Score Category for Uvula/Oropharynx at Day 24 - Pretreatment
Description: as for outcome 9
Time Frame: Day 24 - Pretreatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 27 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

57. Primary Outcome: Percentage of Subjects in Irritation Score Category for Buccal Mucosa at Day 24 - Post-treatment
Description: as for outcome 9
Time Frame: Day 24 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

58. Primary Outcome: Percentage of Subjects in Irritation Score Category for Labial Mucosa at Day 24 - Post-treatment
Description: as for outcome 9
Time Frame: Day 24 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

59. Primary Outcome: Percentage of Subjects in Irritation Score Category for Sublingual Mucosa at Day 24 - Post-treatment
Description: as for outcome 9
Time Frame: Day 24 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

60. Primary Outcome: Percentage of Subjects in Irritation Score Category for Mucobuccal Fold at Day 24 - Post-treatment
Description: as for outcome 9
Time Frame: Day 24 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

61. Primary Outcome: Percentage of Subjects in Irritation Score Category for Gingiva at Day 24 - Post-treatment
Description: as for outcome 9
Time Frame: Day 24 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

62. Primary Outcome: Percentage of Subjects in Irritation Score Category for Tongue at Day 24 - Post-treatment
Description: as for outcome 9
Time Frame: Day 24 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

63. Primary Outcome: Percentage of Subjects in Irritation Score Category for Hard/Soft Palate at Day 24 - Post-treatment
Description: as for outcome 9
Time Frame: Day 24 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

64. Primary Outcome: Percentage of Subjects in Irritation Score Category for Uvula/Oropharynx at Day 24 - Post-treatment
Description: as for outcome 9
Time Frame: Day 24 - Post-treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

65. Primary Outcome: Percentage of Subjects in Irritation Score Category for Buccal Mucosa at Day 25
Description: as for outcome 9
Time Frame: Day 25
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

66. Primary Outcome: Percentage of Subjects in Irritation Score Category for Labial Mucosa at Day 25
Description: as for outcome 9
Time Frame: Day 25
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

67. Primary Outcome: Percentage of Subjects in Irritation Score Category for Sublingual Mucosa at Day 25
Description: as for outcome 9
Time Frame: Day 25
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

68. Primary Outcome: Percentage of Subjects in Irritation Score Category for Mucobuccal Fold at Day 25
Description: as for outcome 9
Time Frame: Day 25
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

69. Primary Outcome: Percentage of Subjects in Irritation Score Category for Gingiva at Day 25
Description: as for outcome 9
Time Frame: Day 25
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

70. Primary Outcome: Percentage of Subjects in Irritation Score Category for Tongue at Day 25
Description: as for outcome 9
Time Frame: Day 25
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

71. Primary Outcome: Percentage of Subjects in Irritation Score Category for Hard/Soft Palate at Day 25
Description: as for outcome 9
Time Frame: Day 25
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

72. Primary Outcome: Percentage of Subjects in Irritation Score Category for Uvula/Oropharynx at Day 25
Description: as for outcome 9
Time Frame: Day 25
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Number analyzed (Participants) | 26 | 26 | 23
Percentage of Participants
  None | 100 | 100 | 100
  Mild | 0 | 0 | 0
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 25, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 8 (Day 25). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | 19292-116-A Control (Listerine®) | 12027-019 | 12027-020
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.